CLINICAL TRIAL: NCT03663517
Title: Gestational Age Specific Thyroid Function Reference Range in Hong Kong
Brief Title: Gestational Age Specific Thyroid Function Reference Range
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Wing Hung Tam, Professor, Chinese University of Hong Kong
Other Study IDs: CUHK_TMP00159
Record Dates: First submitted 2018-08-21; First posted 2018-09-10 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Thyroid; Reference Values; Pregnancy
Keywords: Thyroid; Reference values; Pregnancy
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cord blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pregnant women: pregnant women in Hong Kong

SUMMARY:
It has been well accepted that maternal thyroid dysfunction has adverse affects on both mothers and fetuses. However, the dramatical changes during pregnancy make the interpretation of thyroid function test (TFT, i.e. free triiodothyronine [FT3], free thyroxine [FT4] and thyrotropin [TSH]) very difficult. Previous studies have shown that the level of thyroid hormones differs from non-pregnant population and varies from gestational ages. Moreover, studies have shown the agreement among different instrument platforms was quite low. This study is aimed to determine gestational age specific TFT reference ranges of the local pregnant population for all available platforms currently used under Hospital Authority and Department of Health.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women receiving pregnancy and postnatal care in the Department of Obstetrics & Gynaecology, Prince of Wales Hospital, Hong Kong

Exclusion Criteria:

* 1. Previous history of thyroid dysfunction (hypothyroidism or hyperthyroidism);
* 2. Autoimmune disease, particularly those receiving corticosteroid or immunosuppressant: e.g. systemic lupus erythematosus;
* 3. Disease associated with thyroid dysfunction: e.g. molar pregnancy

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Gestational age-specific thyroid function reference range
Study Population: Hong Kong women
Sampling Method: Probability Sample
Enrollment: 599 (Actual)
Dates: Start 2014-07-02 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2016-04-30 (Actual)

PRIMARY OUTCOMES:
Change of free triiodothyronine (FT3) during pregnancy | At the time of booking for antenatal visit (1st trimester), oral glucose tolerance test (24-32 weeks), admission for delivery (3rd trimester) and a gestational age assigned randomly.
  gestational FT3 level
Change of free thyroxine (FT4) during pregnancy | At the time of booking for antenatal visit (1st trimester), oral glucose tolerance test (24-32 weeks), admission for delivery (3rd trimester) and a gestational age assigned randomly.
  gestational FT4 level
Change of thyrotropin (TSH) during pregnancy | At the time of booking for antenatal visit (1st trimester), oral glucose tolerance test (24-32 weeks), admission for delivery (3rd trimester) and a gestational age assigned randomly.
  gestational TSH level

CONTACTS AND LOCATIONS:
Overall Officials: Wing Hung Tam, MD, Principal Investigator — Chinese University of Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
To be confirmed.